CLINICAL TRIAL: NCT03064581
Title: A Pap Test Intervention to Enhance Decision Making Among Pacific Islander Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California State University, Fullerton (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CSUFR01CA149324; R01CA149324 (NIH)
Record Dates: First submitted 2017-01-12; First posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; Screening; Pap Test; Pacific Islander Americans
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Gender-specific culturally tailored social-support informed educational intervention session.
  Interventions: Behavioral: Intervention
- Control (No Intervention): Usual care with delayed intervention at the end of study.

INTERVENTIONS:
Behavioral: Intervention — The educational session consisted of a one-hour small group discussion (5-10 people). Gender-specific community health educators facilitated sessions for Pacific Islander women and for their spouses/significant others that included an educational video and other materials (brochure, calendar, and resource list). The video emphasized the importance of Pap testing for Pacific Islander women, and showed men supporting their women to get tested. Women's sessions provided basic information on cervical cancer and pap testing, and ended with verbal commitments and target screening dates by women to get screened. The men's education sessions contained similar information, with supplemental information on how to provide support for their wives to get tested and exercises on showing their support.
  Arms: Intervention

SUMMARY:
This community-based randomized trial tested the effects of a social support intervention to increase Chamorro, Samoan, and Tongan women's Pap test behavior and social support among their male spouses or significant others in Southern California.

DETAILED DESCRIPTION:
The purpose of this five-year community-based randomized trial was to: 1) examine the Pap test decision making process in Pacific Islander women; 2) assess the role of social support within the decision making process; and 3) develop and test an intervention to increase Pap testing among Pacific Islander women, and support among their male spouses/significant others. The intervention was created utilizing a Multi-Attribute Utility model and social support theory resulting in gender-specific educational workshops consisting of a social support intervention that informed both Pacific Islander women and men about cervical cancer and the importance of Pap testing for Pacific Islander women, and aimed to increase social support among their male spouses/significant others.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 21 to 65
* Of Chamorro, Samoan, and/or Tongan ethnicity
* Has a significant other (married or in a long-term relationship for more than 5 years).

Exclusion Criteria:

* Not a member of one of the churches or clans visited for recruitment

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1014 (Actual)
Dates: Start 2008-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Change in receipt of a Pap test | Assessed at baseline and 6-month follow-up
  One question regarding whether the woman received a Pap test, among those who had not received one within the past 3 years at baseline

SECONDARY OUTCOMES:
Change in knowledge of cervical cancer risk factors | Assessed at baseline and 6-month follow-up
  Six true/false questions regarding whether risk increases if woman has family history, smokes, has poor hygiene, spouse has many sex partners, had intercourse starting at early age, and has had more than one sex partner
Change in fatalistic attitudes towards cancer | Assessed at baseline and 6-month follow-up
  Five agree/disagree questions regarding whether woman would undergo treatment if diagnosed with cervical cancer, would rather not know if she has cervical cancer, whether she believed there is not much she can do to prevent getting cervical cancer, whether cervical cancer is punishment from god, and whether she would feel less like a woman if she had cervical cancer.
Change in perceived social support | Assessed at baseline and 6-month follow-up
  Fifteen items from the RAND Medical Outcomes Study (MOS) social support survey that use a 4-point likert scale (none, some, a lot, all the time) regarding how much the woman can count on husband to: listen, provide info, give advice, can confide, advice is wanted, can share private worries, will give suggestions, is understanding, can help if bedridden, can take to doctor, can prepare meals, can help with daily chores, shows love, makes women feel wanted, and hugs.
Scheduled a Pap test | Assessed at 6 month follow-up
  Number of women who reported scheduling a Pap test, among women who had not received a Pap test within the past 3 years at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sora Park Tanjasiri, DrPH, Principal Investigator — California State University, Fullerton; Lola Sablan-Santos, Principal Investigator — Guam Communications Network
Locations (1):
- California State University, Fullerton, Fullerton, California, United States

IPD SHARING:
Plan to Share IPD: Yes
After completion of each data collection activity, all program project datasets will be de-identified and then made available for secondary analysis on the California State University, Fullerton, Health Promotion Research Institute website. A consultant, who is experienced in large multi-site controlled trials, will assist with the protocols (in years 2 and 3) required for dataset documentation and distribution. Researchers will be able to access the data, documentation, and surveys by registering on the website, obtaining approval from the Health Promotion Research Institute steering committee, and downloading the files. Care will be taken to ensure that respondents cannot be identified from the information in the public-use dataset. The final dataset will be stripped of identifiers (i.e., individual respondent identifying information, such as names and phone numbers, will be removed) prior to release for sharing.